CLINICAL TRIAL: NCT05273840
Title: Effect of Nutritional Supplements (Ivital Control) on Clinical Outcomes in Patients With Prediabetes and Obesity：a Randomized Controlled Study
Brief Title: Effect of Nutritional Supplements on Clinical Outcomes in Patients With Prediabetes and Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-R037
Record Dates: First submitted 2022-02-10; First posted 2022-03-10 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: PreDiabetes; Obesity
Keywords: PreDiabetes; Obesity; Glycosylated hemoglobin; weight
MeSH Terms: conditions — Prediabetic State; Obesity; Body Weight | interventions — Chocolate

STUDY DESIGN:
Intervention Model Description: 1. life intervention group
  2. nutritional supplement intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- life intervention group (Placebo Comparator): On the basis of the patient's original eating habits, basic dietary and lifestyle guidance is given to the patients until the end of the visit.
  Interventions: Behavioral: lifestyle intervention
- nutritional supplement intervention group (Experimental): On the basis of the patient's original eating habits, basic dietary and lifestyle guidance is given, and at the same time, nutritional supplements(Ivital Control) are given to instead a meal per day. 2 bags once a day until the end of the visit.
  Interventions: Dietary Supplement: Ivital Control

INTERVENTIONS:
Dietary Supplement: Ivital Control — Patients in the intervention group will take 2 sachets of nutritional supplements(Ivital Control) once a day in lieu of one meal, besides receiving lifestyle interventions.
  Other Names: Produced by Fresenius Kabi; Chocolate flavor; Product specifications: 460g (46g*10)
  Arms: nutritional supplement intervention group
Behavioral: lifestyle intervention — Patients will receive lifestyle interventions.
  Arms: life intervention group

SUMMARY:
This study aims to improve blood glucose and weight in patients with prediabetes and obesity through health education, nutritional supplement interventions, clinical evaluation, and close clinical follow-up.100 patients with prediabetes with obesity were randomly divided into 2 groups: life intervention group, nutritional supplement intervention group. All enrolled participants were recommended for routine diabetes lifestyle education according to the "Expert Consensus on Prediabetes Intervention in Adults in China". The duration of the intervention was 3 months. The investigators aimed to compare the differences in weight, glycosylated hemoglobin, lipids and other indicators of the two groups of included populations before and after the intervention. In addition, the investigators are to explore the effects of nutritional supplement interventions on glycolipid metabolism and body weight in prediabetes with obesity.

ELIGIBILITY:
Inclusion Criteria:

* According to the American Diabetes Society (ADA) 2010 standard: meet one of the following (1) fasting blood glucose at 100 mg/dl to 125 mg/dl; (2) sugar load 2h blood glucose at 140 mg/dl to 199 mg/dl; (3) glycosylated hemoglobin in 5.7% to 6.4%
* Body mass index (BMI) ≥ 25 and ≤ 35kg/m2
* Have lived locally for at least half a year and have a fixed residence
* No other clinical trials were participated in in the 3 months prior to the trial
* Mental health, being able to take care of oneself in life

Exclusion Criteria:

* People with confirmed diabetes
* Weight change of more than 10% over the past 3 months
* Pregnant or lactating women, men and women planning to become pregnant within two years, or unwilling and unable to use contraception during the study period (women only)
* People who are allergic to the ingredients of nutritional supplements
* Those who have lost weight by any medication (including appetite suppressants such as fluprophenylpropanine, progesterone, laxatives, etc., and diet pills with various Traditional Chinese medicine ingredients) or surgery in the past 3 months
* Patients who have received medical treatment for the following diseases in the past 3 months: diabetes, cholecystitis, peptic ulcer, inflammatory bowel disease, acute urinary tract infection, hyperthyroidism, etc., or patients with chronic gastrointestinal diseases with symptoms of nausea, vomiting and diarrhea in the past month
* Suffer from severe organic diseases such as cancer, coronary heart disease, myocardial infarction and stroke
* Presence of pituitary-adrenal axis dysfunction; secondary obesity due to other diseases (e.g., Cushing syndrome, hypothyroidism, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
the proportions of participants regressing back to normal glucose level | 3 months
  The normal glucose level was defined as FPG < 6.1 mmol/L and 2hPG < 7.8 mmol/L during the OGTT.

SECONDARY OUTCOMES:
change in HbA1c | 3 months
  change in HbA1c
body weight | 3 months
  changes in body weight

OTHER OUTCOMES:
changes in waist circumference | 3 months
  anthropometric parameters
changes in hip circumference | 3 months
  anthropometric parameters
changes in neck circumference | 3 months
  anthropometric parameters
changes in visceral fat area | 3 months
  body composition
changes in body fat percentage | 3 months
  body composition
changes in lean mass | 3 months
  body composition
blood lipids | 3 months
  changes in LDL-cholesterol, HDL-cholesterol
changes in triglyceride level (blood lipids) | 3 months
  changes in triglyceride

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, China

IPD SHARING:
Plan to Share IPD: No